CLINICAL TRIAL: NCT05386160
Title: Department of Ophthalmology, Ruijin Hospital, Affiliated Medical School, Shanghai Jiaotong University
Brief Title: Phacoemulsification Combined With Intravitreal Injection of Ranibizumab Prevent Postoperative Capillary Non-perfusion Zone Progress in Non-proliferative Diabetic Retinopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RuijinH202201
Record Dates: First submitted 2022-04-26; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-01

CONDITIONS: Mild Non-proliferative Diabetic Retinopathy; Cataract Diabetic; Diabetic Retinopathy
Keywords: Phaco; VEGF; diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab; Phacoemulsification

STUDY DESIGN:
Intervention Model Description: This research is a single-center prospective, randomized controlled study. Patient were divided into two groups, the control group is phacoemulsification surgery group and the intervention group is phacoemulsification surgery combine intravitreal injection of Ranibizumab group.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cataract phacoemulsification combines Ranibizumab (Active Comparator): 0.05 ml of ranibizumab was injected into the vitreous immediately after the operation
  Interventions: Drug: Ranibizumab Injection [Lucentis]
- Cataract phacoemulsification (Active Comparator): 0.05 ml of ranibizumab was injected into the vitreous immediately after the operation
  Interventions: Drug: Ranibizumab Injection [Lucentis]; Device: Phacoemulsification

INTERVENTIONS:
Drug: Ranibizumab Injection [Lucentis] — intravitreal injection of Ranibizumab；
  Other Names: Phacoemulsification
Device: Phacoemulsification — Phacoemulsification
  Arms: Cataract phacoemulsification

SUMMARY:
Diabetic retinopathy has been found progress in 20-70% diabetic patient after cataract phacoemulsification surgery. Intravitreal injection of anti-VEGF Ranibizumab is an important treatment for diabetic retinopathy including non-proliferative diabetic retinopathy (NPDR). However, there is no research about phacoemulsification surgery combine Intravitreal injection of Ranibizumab on diabetic retinopathy. The research focus on the effect of phacoemulsification surgery combine intravitreal injection of Ranibizumab on mild non-proliferative diabetic retinopathy and explore the reasons for differences in treatment outcomes.

DETAILED DESCRIPTION:
This research is a single-center prospective, randomized controlled study. Patient were divided into two groups, the control group is phacoemulsification surgery group and the intervention group is phacoemulsification surgery combine intravitreal injection of Ranibizumab group. Eye examination including visual acuity, intraocular pressure(IOP), fundus fluoroscopy, macular optical coherence tomograph（OCT） examination, were taken before cataract surgery. The anterior aqueous humor was extracted before cataract phacoemulsification in the combined operation group, and 0.05 ml of ranibizumab was injected into the vitreous immediately after the operation. The aqueous humor concentrations of vascular endothelial growth factor（VEGF）, interleukin（IL）IL-2, IL-4, and Tumor Necrosis Factor（TNF） were checked by real-time polymerase chain reaction assay（RT-PCR） and ELISA analysis. The Best Corrected Visual Acuity（BCVA）, IOP and fundus lesions changes were observed in the two groups after operation. Diabetic retinopathy capillary non-perfusion zone were evaluated one year after phacoemulsification surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Commitment to follow the research procedures and cooperate with the implementation of the whole process of research
* No specific gender, 18+ years old
* Diagnosed in line with NPDR,
* Phacoemulsification combined with anti-VEGF therapy is planned
* No obvious surgical contraindications

Exclusion Criteria:

* Use of other investigational drug treatments or take part in other types of clinical studies
* Allergy to anti-VEGF drugs
* Patients with other macular and optic disc diseases
* Patients with meaningful diabetic macular edema
* Patient with surgical complications

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
capillary non-perfusion zone of non-proliferative diabetic retinopathy | 1 year
  Patient were divided into two groups, the control group is phacoemulsification surgery group and the intervention group is phacoemulsification surgery combine intravitreal injection of Ranibizumab group. Eye examination including visual acuity, intraocular pressure (IOP), fundus fluoroscopy, macular OCT examination, were taken before cataract surgery. The anterior aqueous humor was extracted before cataract phacoemulsification in the combined operation group, and 0.05 ml of ranibizumab was injected into the vitreous immediately after the operation. The BCVA, IOP and fundus lesions changes were observed in the two groups after operation. Diabetic retinopathy capillary non-perfusion zone were evaluated one year after phacoemulsification surgery.

SECONDARY OUTCOMES:
Determination of inflammatory factors in anterior aqueous humor | before cataract phacoemulsification
  The anterior aqueous humor was extracted before cataract phacoemulsification in the combined operation group. The aqueous humor concentrations of VEGF, IL-2, IL-4, and TNF were checked by RT-PCR and ELISA analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zijian Yang, Dr, Study Director — Department of Ophthalmology, Ruijin Hospital north, Affiliated Medical School, Shanghai Jiaotong University
Locations (1):
- Department of Ophthalmology, Ruijin Hospital Affiliated Medical,Shanghai Jiaotong University School, Shanghai, Shanghai Municipality, China